CLINICAL TRIAL: NCT05556369
Title: Genetic Characterization of Cardiomyopathies (POLICARDIOMIO2021)
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Stefano Carugo, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 2385
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cardiomyopathies
Keywords: Cardiomyopathy; Hypertrophic; Dilated; ARVD; Restrictive; NGS; Gene mutation
MeSH Terms: conditions — Cardiomyopathies; Hypertrophy; Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm Study: The study involves the execution of a genetic analysis using a panel of 54 genes conducted on blood obtained from peripheral venous sampling, the collection of clinical / instrumental / biological data in a dedicated prospective register in the form of a pseudo-anonymized database and the follow-up clinical up over time of patients. The study also provides for the execution of: a cardiological examination with electrocardiogram, Echocardiogram-color doppler and Basic blood tests: CBC, renal function, electrolytes, hepatic profile, NT-proBNP, lipid profile.

SUMMARY:
Cardiomyopathy refers to a diverse group of myocardial diseases with multiple causes. In 1995, the World Health Organization classified cardiomyopathies into hypertrophic, dilated, restrictive, and mixed type. This classification is based on the pathophysiology of the disease. However, with rapid evolution of molecular genetics in cardiology, the American Heart Association in 2006 has classified cardiomyopathies into two major groups based on predominant organ involvement and etiology; Primary cardiomyopathies are those solely or predominantly confined to heart muscle and are relatively few in number. Secondary cardiomyopathies show pathologic myocardial involvement as part of a large number and variety of generalized systemic (multiorgan) disorders.Current evidence supports the use of genetic testing in clinical practice to improve risk stratification for clinically affected patients and their at-risk relatives for cardiomyopathies.

ELIGIBILITY:
Inclusion Criteria:

* Presence of structural cardiomyopathy
* First degree relatives for cardiomyopathy

Exclusion Criteria:

* Age > 80
* Presence of sufficient conditions to explain the clinical condition of cardiomyopathy
* Peripartum cardiomyopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referred to Cardiology Department of Policlinico di Milano for the diagnosis of suspicious Cardiomyopathy or First degree relatives for cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Genetic Characterization | 5 years
  To perform a genetic characterization of subjects affected by structural cardiomyopathies with clinical suspicion of genetic pattern

SECONDARY OUTCOMES:
Genetic and phenotypic characterization of the first degree relatives | 5 years
  To perform a genetic and phenotypic characterization of the first degree relatives of a subject affected by genetic structural cardiomyopathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Lombardy, Italy